CLINICAL TRIAL: NCT04004663
Title: A PHASE 1, RANDOMIZED, OPEN-LABEL, CROSS-OVER, SINGLE DOSE STUDY TO ESTIMATE THE RELATIVE BIOAVAILABILITY OF CANDIDATE CAPSULE FORMULATIONS OF PF-06651600 RELATIVE TO TABLETS IN HEALTHY PARTICIPANTS
Brief Title: Bioavailability Study of PF-06651600 Formulations in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B7981022; 2019-001452-19 (EudraCT Number)
Record Dates: First submitted 2019-06-28; First posted 2019-07-02 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Healthy Volunteers
Keywords: pharmacokinetics; JAK inhibitor; PF-06651600
MeSH Terms: interventions — PF-06651600

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Treatment Sequence 1 (Experimental): Participants will receive a single dose of each formulation of PF-06651600 in each period as follows: Period 1 (Treatment A); Period 2 (Treatment B); Period 3 (Treatment C); Period 4 (Treatment D).
  Interventions: Drug: PF-06651600
- Treatment Sequence 2 (Experimental): Participants will receive a single dose of each formulation of PF-06651600 in each period as follows: Period 1 (Treatment B); Period 2 (Treatment D); Period 3 (Treatment A); Period 4 (Treatment C).
  Interventions: Drug: PF-06651600
- Treatment Sequence 3 (Experimental): Participants will receive a single dose of each formulation of PF-06651600 in each period as follows: Period 1 (Treatment C); Period 2 (Treatment A); Period 3 (Treatment D); Period 4 (Treatment B).
  Interventions: Drug: PF-06651600
- Treatment Sequence 4 (Experimental): Participants will receive a single dose of each formulation of PF-06651600 in each period as follows: Period 1 (Treatment D); Period 2 (Treatment C); Period 3 (Treatment B); Period 4 (Treatment A).
  Interventions: Drug: PF-06651600

INTERVENTIONS:
Drug: PF-06651600 — PF-06651600 100 milligrams (mg) will be provided in 4 different oral formulations (Treatment A,B,C,D). Participants will receive each formulation in one of 4 periods

SUMMARY:
The study will be conducted as a Phase 1, open-label, single dose, randomized, 4-period, cross over design in a single cohort of approximately 12 healthy male or female participants at a single center. Participants will be randomized into 1 of 4 sequences of treatment.

ELIGIBILITY:
INCLUSION CRITERIA:

* Participants who are healthy as determined by medical evaluation including a detailed medical history, complete physical examination, which includes BP and pulse rate measurement, clinical laboratory tests, and 12 lead ECG.
* Participants with body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).

EXCLUSION CRITERIA

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, dermatological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
* Known immunodeficiency disorder, including positive serology for human immunodeficiency virus (HIV) at screening, or a first degree relative with a hereditary immunodeficiency.
* Infection with hepatitis B or hepatitis C viruses

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time profile from time zero extrapolated to infinite time (AUCinf)of PF-06651600 | Day 1 pre-dose and at 0.25, 0.5, 1, 2, 3, 4, 6, 12, and 16 hrs, and Day 2, at 24 hours post-dose in Periods 1-4.
Maximum plasma PF-06651600 concentration (C max) | Day 1 pre-dose and at 0.25, 0.5, 1, 2, 3, 4, 6, 12, and 16 hrs, and Day 2, at 24 hours post-dose in Periods 1-4.

SECONDARY OUTCOMES:
Single dose time to reach maximum observed plasma concentration (Tmax) of PF-06651600 | Day 1 pre-dose and at 0.25, 0.5, 1, 2, 3, 4, 6, 12, and 16 hrs, and Day 2, at 24 hours post-dose in Periods 1-4.
Single dose Area under the Curve from Time Zero to Last quantifiable concentration [AUC last) of PF-06651600 | Day 1 pre-dose and at 0.25, 0.5, 1, 2, 3, 4, 6, 12, and 16 hrs, and Day 2, at 24 hours post-dose in Periods 1-4.
Single dose plasma decay half-life (t 1/2) of PF-06651600 | Day 1 pre-dose and at 0.25, 0.5, 1, 2, 3, 4, 6, 12, and 16 hrs, and Day 2, at 24 hours post-dose in Periods 1-4.
Single dose Apparent Oral Clearance (CL/F) of PF-06651600 | Day 1 pre-dose and at 0.25, 0.5, 1, 2, 3, 4, 6, 12, and 16 hrs, and Day 2, at 24 hours post-dose in Periods 1-4.
Single dose Apparent Volume of Distribution (Vz/F) of PF-06651600 | Day 1 pre-dose and at 0.25, 0.5, 1, 2, 3, 4, 6, 12, and 16 hrs, and Day 2, at 24 hours post-dose in Periods 1-4.
Frequency of abnormal safety laboratory tests | Baseline up to day 9
Frequency of Adverse Events | Baseline up to Day 35

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Brussels Clinical Research Unit, Brussels, Be-bru, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Saadeddin A, Purohit V, Huh Y, Wong M, Maulny A, Dowty ME, Sagawa K. Virtual Bioequivalence Assessment of Ritlecitinib Capsules with Incorporation of Observed Clinical Variability Using a Physiologically Based Pharmacokinetic Model. AAPS J. 2024 Jan 24;26(1):17. doi: 10.1208/s12248-024-00888-9. PMID 38267790
- [Derived] Wojciechowski J, S Purohit V, Huh Y, Banfield C, Nicholas T. Evolution of Ritlecitinib Population Pharmacokinetic Models During Clinical Drug Development. Clin Pharmacokinet. 2023 Dec;62(12):1765-1779. doi: 10.1007/s40262-023-01318-3. Epub 2023 Nov 2. PMID 37917289
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981022